CLINICAL TRIAL: NCT02351713
Title: Is a Threshold-Based Model a Superior Method to the Relative Percent Concept for Establishing Individual Exercise Intensity? A Randomized Controlled Trial
Brief Title: Comparison of Exercise Intensity Prescription
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Western Colorado University (Other)
Responsible Party: Principal Investigator, Lance Dalleck, Assistant Professor, Western Colorado University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WesternSCU
Record Dates: First submitted 2015-01-22; First posted 2015-01-30 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Cardiovascular Disease
Keywords: primary prevention
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Threshold based method (Experimental): Exercise Week 1 Heart rate (HR) < first ventilatory threshold (VT1) 3 days 20 min/day Week 2 HR < VT1 4 days 25 min/day Week 3 HR < VT1 4 days 30 min/day Week 4 HR < VT1 5 days 30 min/day Week 5-6 HR ≥ VT1 to < second ventilatory threshold (VT2) 5 days 30 min/day Weeks 7-8 HR ≥ VT1 to < VT2 5 days 30 min/day Weeks 9-12 HR ≥ VT2 5 days 30 min/day
  Interventions: Other: Exercise
- Relative percent method (Experimental): Exercise Week 1 40-45% heart rate reserve 3 days 20 min/day Week 2 40-45% heart rate reserve 4 days 25 min/day Week 3 40-45% heart rate reserve 4 days 30 min/day Week 4 40-45% heart rate reserve 5 days 30 min/day Week 5-6 50-55% heart rate reserve 5 days 30 min/day Weeks 7-8 50-55% heart rate reserve 5 days 30min/day Weeks 9-12 60-65% heart rate reserve 5 days 30 min/day
  Interventions: Other: Exercise
- Control (No Intervention): Non-exercise control group

INTERVENTIONS:
Other: Exercise — Continuous aerobic exercise prescribed according to two exercise intensity methods: threshold based method (i.e., ventilatory threshold) and relative percent method (i.e., heart rate reserve).
  Arms: Relative percent method; Threshold based method

SUMMARY:
Therefore, the purpose of this study is to compare the effectiveness of two exercise training programs for improving cardiorespiratory fitness: the ACE three-zone training model (i.e., threshold based training) versus the more common ACSM recommended relative percent method (i.e., %HRR).

It is hypothesized that:

1. The ACE three-zone training model will elicit greater mean changes in cardiorespiratory fitness (as measured by VO2max) when compared to the relative percent method.
2. Participants in the ACE three-zone training model group will be more likely to have favorable VO2max responses; while comparatively, participants in the relative percent method group would be more likely to experience a VO2max nonresponse to exercise training.

DETAILED DESCRIPTION:
Cardiorespiratory fitness, typically determined by maximal oxygen uptake (VO2max), is a fundamental measurement for the exercise physiologist and other health professionals. VO2max refers to the highest rate at which oxygen can be taken up and consumed by the body during intense exercise. The "F.I.T.T." principle is an acronym for the four components for exercise prescription: frequency, intensity, time (length), and type of exercise.

Exercise intensity is arguably the most critical component of the exercise prescription model. Failure to meet minimal threshold values may result in lack of a training effect, while too high of an exercise intensity could lead to over-training and negatively impact adherence to an exercise program. The traditional reference standard for prescribing exercise intensity is expressed in terms of percentages of heart rate reserve (%HRR) or oxygen uptake reserve (%VO2R). This is considered the 'relative percent method'. The American College of Sports Medicine (ACSM) currently recommends an exercise intensity of 40-59% HRR/VO2R for improving and maintaining cardiorespiratory fitness. Nevertheless, despite a large evidence base supporting the ACSM relative percent concept recommendation for prescribing exercise intensity, there is concern that the approach consists of a very large range of acceptable percentages and fails to take into account individual metabolic responses to exercises. This study sought to compare the effectiveness of two exercise training programs for improving cardiorespiratory fitness: the ACE three-zone training model (i.e., threshold based training) versus the more common ACSM recommended relative percent concept (i.e., %HRR).

Apparently healthy, but sedentary men and women (n = 42) were randomized to a non-exercise control group or one of two exercise training groups. Exercise training was performed 30 min/day on 5 days/wk for 12wk according to one of two exercise intensity regimens: 1) a relative percent method was used in which intensity was prescribed according to percentages of heart rate reserve (HRR group), or 2) a threshold based method (ACE-3ZM) was used in which intensity was prescribed according to the first ventilatory threshold (VT1) and second ventilatory threshold (VT2).

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for inclusion into the study if they were low-to-moderate risk as defined by the ACSM and sedentary.
* Participants were also eligible for inclusion into the study if they verbally agreed to continue previous dietary habits and not perform additional exercise beyond that required for the present study.

Exclusion Criteria:

* Exclusionary criteria included evidence of cardiovascular pulmonary, and/or metabolic disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2max) as a measure of cardiorespiratory fitness | 12 weeks
Estimate of 10-year Cardiovascular Disease Risk | 12 weeks

REFERENCES:
- [Derived] Wolpern AE, Burgos DJ, Janot JM, Dalleck LC. Is a threshold-based model a superior method to the relative percent concept for establishing individual exercise intensity? a randomized controlled trial. BMC Sports Sci Med Rehabil. 2015 Jul 4;7:16. doi: 10.1186/s13102-015-0011-z. eCollection 2015. PMID 26146564